CLINICAL TRIAL: NCT01304212
Title: Comparison of the Analgesic Effect of Femoral Nerve Block, Intraarticular Infiltration or a Combination of Both in the Control of Pain in Total Knee Arthroplasty
Brief Title: Effectiveness of Analgesia in Total Knee Arthroplasty
Acronym: ATR-2011
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jose Antonio Bernia Gil (Other)
Responsible Party: Sponsor-Investigator, Jose Antonio Bernia Gil, PhD,MD, Consorci Sanitari de Terrassa
Organization: Consorci Sanitari de Terrassa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATR-2011
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Pain
Keywords: total knee arthroplasty; intraarticular infiltration; femoral block
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- femoral block (Active Comparator)
  Interventions: Drug: ropivacaine
- local infiltration + femoral nerve block (Experimental): Combination of local infiltration with drugs and femoral nerve block
  Interventions: Drug: morphine ,ketorolac
- several drugs local infiltration (Active Comparator)
  Interventions: Drug: several drugs: morphine chloride,ropivacaine,epinephrine,ketorolac; Drug: ropivacaine,morphine chloride,epinephrine,ketorolac

INTERVENTIONS:
Drug: several drugs: morphine chloride,ropivacaine,epinephrine,ketorolac — This technique is performed intraoperatively with a 100 ml solution containing: 225 mg of ropivacaine 1% (22.5 ml) + 5 mg of morphine chloride 0.1% (5ml) + 30 mg of epinephrine 1:1000 (0.3 ml ) + ketorolac 30mg (1ml) +71 ml of 0.9% saline
  Arms: several drugs local infiltration
Drug: ropivacaine,morphine chloride,epinephrine,ketorolac — This technique is performed intraoperatively with a 100 ml solution containing: 225 mg of ropivacaine 1% (22.5 ml) + 5 mg of morphine chloride 0.1% (5ml) + 30 mg of epinephrine 1:1000 (0.3 ml ) + ketorolac 30mg (1ml) +71 ml of 0.9% saline
  Arms: several drugs local infiltration
Drug: ropivacaine — The lock is held before starting the operation, viewing with ultrasound and confirmed the femoral nerve with nerve stimulation at an intensity of 0.5 mA and a frequency of 2 Hz Pajunk 50mm needle, patellar flexion. It be administered 30ml of ropivacaine 0.75% (225mg)
  Arms: femoral block
Drug: morphine ,ketorolac — ultrasound-assisted femoral nerve block is performed and leaks intraoperatively with a 100 ml solution containing: 5 mg of morphine to 0.1% (5ml) +30 mg of ketorolac (1 ml) +96 ml of 0.9% saline.
  Arms: local infiltration + femoral nerve block

SUMMARY:
The purpose of this study is to compare the analgesic effectiveness of three techniques: the femoral nerve block, intraarticular infiltration or a combination of both in the control of pain in total knee arthroplasty (KA). The hypothesis to be tested in this study is that the performance multimodal postoperative pain KA combining two analgesic techniques to obtain better analgesia than when applied separately.

ELIGIBILITY:
Inclusion Criteria:

* intervention program for total knee arthroplasty
* ASA I, II, III
* over 65 years old

Exclusion Criteria:

* ASA > III
* patients who refuse the realization of technical loco-regional anesthesia
* presence of coagulopathy or impaired hemostatic function
* BMI > 35
* Serious intraoperative complications
* patients undergoing bypass and aortic-femoral or femoro popliteal bypass operated leg
* patients treated for chronic pain diagnosed processes, different knee osteoarthritis

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 48 hours postoperatively
  Is measured at the time of starting rehabilitation, postoperatively 48 hours using visual analog scale, numerical and categorical verbal pain scale at 12,24 and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Bernia Gil, MD, PhD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain